CLINICAL TRIAL: NCT00047307
Title: A Phase 1 Study of Alvocidib (Flavopiridol) in Combination With Radiation in Locally Advanced, Non-Operable Pancreatic and Extrahepatic Bile Duct Cancers
Brief Title: Flavopiridol Plus Radiation Therapy Followed By Gemcitabine Hydrochloride in Treating Patients With Locally Advanced, Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01430; 02-057; NCI-5764; MSKCC-02057; CDR0000257662; U01CA069856 (NIH); R01CA067819 (NIH)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — alvocidib; Gemcitabine; Radiotherapy, Conformal

ARMS (1):
- Treatment (alvocidib, gemcitabine hydrochloride, 3DRT) (Experimental): Patients receive flavopiridol IV over 1 hour twice weekly (on days 1 and 4 or days 2 and 5) for 6 weeks. Concurrently, patients undergo radiotherapy once daily 5 days a week for 5.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Four weeks after the completion of radiotherapy, patients are re-evaluated*. Beginning within 4-7 weeks after the completion of chemotherapy and radiotherapy, patients receive gemcitabine hydrochloride alone or in combination with another cytotoxic agent or gemcitabine hydrochloride combined with a targeted drug (e.g., erlotinib or bevacizumab) at the discretion of the oncologist. NOTE: *Patients whose imaging studies suggest potential curative resection are referred for a surgical evaluation before initiating gemcitabine hydrochloride therapy. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. Continued (see detailed description)
  Interventions: Drug: alvocidib; Drug: gemcitabine hydrochloride; Radiation: 3-dimensional conformal radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Radiation: 3-dimensional conformal radiation therapy — Undergo 3-dimensional conformal radiation therapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy work different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Flavopiridol may make the tumor cells more sensitive to radiation therapy. Phase I trial to study the effectiveness of combining flavopiridol with radiation therapy followed by gemcitabine hydrochloride in treating patients who have locally advanced, unresectable pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of flavopiridol in combination with radiotherapy followed by gemcitabine in patients with locally advanced, unresectable pancreatic cancer.

II. Determine the toxicity of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of flavopiridol in these patients. II. Determine, preliminarily, the therapeutic activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of flavopiridol.

Patients receive flavopiridol IV over 1 hour twice weekly (on days 1 and 4 or days 2 and 5) for 6 weeks. Concurrently, patients undergo radiotherapy once daily 5 days a week for 5.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Four weeks after the completion of radiotherapy, patients are re-evaluated*. Beginning within 4-7 weeks after the completion of chemotherapy and radiotherapy, patients receive gemcitabine hydrochloride alone or in combination with another cytotoxic agent or gemcitabine hydrochloride combined with a targeted drug (e.g., erlotinib or bevacizumab) at the discretion of the oncologist. NOTE: *Patients whose imaging studies suggest potential curative resection are referred for a surgical evaluation before initiating gemcitabine hydrochloride therapy. Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are treated at the recommended phase II dose.

Patients are followed at 4 weeks and then every 8 weeks thereafter.

PROJECTED ACCRUAL: Approximately 3-46 patients will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * No non-adenocarcinoma of the pancreas (i.e., islet cell, lymphoma, or sarcoma)
  * Locally advanced and unresectable disease defined as the following:

    * Obvious encasement of the celiac, hepatic, or superior mesenteric artery
    * Encasement of the portal or superior mesenteric vein not amenable to resection
    * Extrapancreatic extension with or without regional lymph node involvement
    * No distant metastases
* Measurable or evaluable disease

  * Primary pancreatic tumor is considered evaluable, not measurable
  * A lymph node mass is considered measurable
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No Crohn's disease or inflammatory bowel disease that would preclude study participation
* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
* No other uncontrolled concurrent illness that would preclude study participation
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior chemotherapy for this disease except gemcitabine hydrochloride-based therapy for which no radiologic evidence of distant metastatic disease exists
* No prior flavopiridol or other cyclin-dependent kinase therapies
* No prior radiotherapy for this disease
* Prior curative surgery with local recurrence allowed
* No other concurrent investigational therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2002-08; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of flavopiridol when administered biweekly in conjunction with radiation for patients with locally advanced pancreatic or extrahepatic bile duct cancer | 6 weeks

SECONDARY OUTCOMES:
Molecular correlates of apoptosis including PARP cleavage and caspase-3 activation, as well as changes in expression of p21, phosphorylation status of pRb and cyclin D1 | Baseline
  Will be summarized by descriptive statistics and used to generate hypothesis for further studies.
Molecular correlates of apoptosis including PARP cleavage and caspase-3 activation, as well as changes in expression of p21, phosphorylation status of pRb and cyclin D1 | 10 weeks
  Will be summarized by descriptive statistics and used to generate hypothesis for further studies.

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States